CLINICAL TRIAL: NCT01963000
Title: Reduction of Mortality in Community-Acquired Pneumonia After Implementing Standardized Care Bundles in the Emergency Department
Brief Title: Standardized Emergency Care for Community Acquired Pneumonia (CAP)
Status: Completed | Type: Observational
Sponsor: Klinikum Nürnberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Christ, Prof. Dr. med. Michael Christ, Klinikum Nürnberg
Other Study IDs: CAP01ED
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Community Acquired Pneumonia; Pneumonia; Infection
Keywords: Community Acquired Pneumonia; Emergency Department; Standardized Care; Reduced Mortality; CRB-65 Risk Classes; Antibiotic Therapy
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia; Infections; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CAP: A patient with CAP was identified by encoding pneumonia without severe immunosuppression (HIV infection, solid organ or bone marrow/stem cell transplants, severe neutropenia) as the main diagnosis (ICD 10 GM) of hospital admission.

SUMMARY:
Community acquired pneumonia (CAP) is associated with a high in-hospital mortality. Standardization of diagnostics and adherence to sepsis bundles in the emergency department (ED) are associated with reduced mortality in patients with sepsis. Investigators examined whether the introduction of standardized care bundles and check lists in the ED are associated with a reduced mortality rate in patients hospitalized for CAP.

This is an observational trial. The investigators retrospectively analyzed performance indicators of 2819 consecutive patients with CAP admitted to the Nuremberg Hospital, Germany, from 2008 to 2009. At the turn of the year, implementation of CAP care bundles took place including interprofessional education, checklists and institutionalized feedback. Primary endpoint was in-hospital mortality of CAP patients. After the implementation of CAP care bundles in the ED, mortality of affected patients was significantly lower in 2009 compared to 2008. This study should demonstrate that the implementation of a standardized CAP care bundle in the ED is associated with a risk reduction in affected patients. Standardization of diagnostic and therapeutic processes in the ED therefore improves the outcome of patients hospitalized for CAP.

ELIGIBILITY:
Inclusion Criteria:

* all patients with community acquired pneumonia

Exclusion Criteria:

* exacerbation of chronic obstructive pulmonary disease
* malignancy
* immunosuppression
* neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department patients
Sampling Method: Probability Sample
Enrollment: 2819 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
mortality of CAP patients | up to 14days

SECONDARY OUTCOMES:
mortality up to 14days in subgroups | up to 14 days
  Mortality of patients upt to 14day is determined in subgroups (different age groups, sub-groups of CRB-risk classes)
  CRB-65: C mental confusion; R respiratory rate ≥30/min; B systolic blood pressure <90 mm Hg; 65, age ≥65 years

CONTACTS AND LOCATIONS:
Locations (1):
- City Hospital Nuremberg, Nuremberg, Bavaria, Germany